CLINICAL TRIAL: NCT02461147
Title: Initial Cholecystectomy With Intraoperative Cholangiography for Patients at Intermediate Risk of Common Bile Duct Stone Migration : Prospective Validation and Analysis
Brief Title: Prospective Validation of "Cholecystectomy First" Strategy for Gallstone Migration
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Pouya Iranmanesh, MD, University Hospital, Geneva
Other Study IDs: CCK first validation
Record Dates: First submitted 2015-01-19; First posted 2015-06-03 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Choledocholithiasis; Gallstone Migration; Cholecystitis; Gallstone Pancreatitis; Cholangitis
MeSH Terms: conditions — Choledocholithiasis; Cholecystitis; Cholangitis | interventions — Cholecystectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Validation cohort: All patients of the study (single group, single arm) will undergo initial cholecystectomy with intraoperative cholangiogram, followed if required by ERCP, according to the standard protocol of treatment previously implemented at the investigators institution.
  Interventions: Procedure: Cholecystectomy with intraoperative cholangiogram

INTERVENTIONS:
Procedure: Cholecystectomy with intraoperative cholangiogram — cf. arm/group description. This intervention is not assigned by the investigators: it is the standard treatment at the investigators institution.

SUMMARY:
Initial cholecystectomy with intraoperative cholangiogram, followed if required by ERCP, has been implemented at the investigators institution as the standard management strategy for patients at intermediate risk of common bile duct stone migration, following a randomized controlled trial previously published by the same investigators team. The aim of this study is to prospectively analyze the outcomes of this strategy.

DETAILED DESCRIPTION:
A previous randomized controlled trial comparing initial cholecystectomy with intraoperative cholangiogram (IOC) versus common bile duct (CBD) assessment and subsequent cholecystectomy for patients admitted in the emergency room with an acute gallstone-related condition and with an intermediate risk of common bile duct stone was performed by the investigators. This study had been registered on Clinicaltrials.gov as well and had shown that a strategy with initial cholecystectomy significantly decreased the length of hospital stay and the number of CBD investigations procedures.

Initial cholecystectomy with IOC is now the standard management strategy for these patients in the investigators hospital. The goal of this study is to perform a prospective validation of this strategy and to analyze if the results obtained in the previously mentioned randomized controlled trial are confirmed on a larger patients cohort. This study will be observational, since the intervention (initial cholecystectomy) is not assigned by the investigators, but is already a standard treatment strategy at our institution.

ELIGIBILITY:
Inclusion Criteria:

* Admission through emergency department for an acute gallstone-related condition (cholecystitis, gallstone pancreatitis, ascending cholangitis, suspicion of gallstone migration, choledocholithiasis)

Exclusion Criteria:

* Severe sepsis or septic shock
* contra-indication to surgery
* previous surgery interfering with common bile duct assessment procedures (roux-en-y gastric bypass, etc.)
* previous cholecystectomy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients admitted through the emergency department for an acute gallstone-related condition.
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2013-09; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay [days] | 1-100 days

SECONDARY OUTCOMES:
Number of common bile duct investigations [N] | Anytime during hospital stay, an expected average of 7 days
  These include number of endoscopic ultrasounds (EUS), magnetic cholangio-pancreatography (MRCP) and endoscopic retrograde cholangio-pancreatography (ERCP) performed during the patient's hospital stay
Common bile duct clearance rate [%] | This outcome will be assessed after each ERCP performed during hospital stay, an expected average of 7 days
  Percentage of patients where common bile duct (CBD) clearance was achieved after ERCP (did not require surgical exploration because of ERCP failure)
Morbidity | From admission up to 6 months after hospital discharge
  Morbidity will be assessed for each patient according to the Dindo-Clavien classification of surgical complications, including death.

CONTACTS AND LOCATIONS:
Overall Officials: Pouya Iranmanesh, MD, Principal Investigator — Geneva University Hospital, Division of Digestive Surgery; Christian Toso, MD-PhD, Study Director — Geneva University Hospital, Division of Digestive Surgery
Locations (1):
- Geneva University Hospital, Geneva, Switzerland

REFERENCES:
- [Result] Iranmanesh P, Frossard JL, Mugnier-Konrad B, Morel P, Majno P, Nguyen-Tang T, Berney T, Mentha G, Toso C. Initial cholecystectomy vs sequential common duct endoscopic assessment and subsequent cholecystectomy for suspected gallstone migration: a randomized clinical trial. JAMA. 2014 Jul;312(2):137-44. doi: 10.1001/jama.2014.7587. PMID 25005650
- [Result] Iranmanesh P, Frossard JL, Toso C. Treatment for patients at intermediate risk of a common duct stone--reply. JAMA. 2014 Nov 19;312(19):2043-4. doi: 10.1001/jama.2014.13425. No abstract available. PMID 25399287
- [Result] Iranmanesh P, Frossard JL, Toso C. Reply: To PMID 25451658. Gastroenterology. 2015 Jan;148(1):252. doi: 10.1053/j.gastro.2014.11.016. Epub 2014 Nov 21. No abstract available. PMID 25451659